CLINICAL TRIAL: NCT01850888
Title: 131I-Metaiodobenzylguanidine (131I-MIBG) Therapy for Refractory Neuroblastoma and Pheochromocytoma
Brief Title: MIBG for Refractory Neuroblastoma and Pheochromocytoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012LS107
Record Dates: First submitted 2013-03-26; First posted 2013-05-10 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Relapsed Neuroblastoma; Metastatic Pheochromocytoma
Keywords: neuroblastoma; pheochromocytoma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma | interventions — 3-Iodobenzylguanidine; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131 I-MIBG Treatment Arm (Experimental): Therapeutic 131 I-Metaiodobenzylguanidine (131I-MIBG) will be infused intravenously, intravenous fluids will be administered to help maintain urine flow and isotope excretion. Potassium iodide solution will be administered to protect thyroid function. G-CSF will be used if necessary for neutrophil recovery. Hematopoietic stem cell infusion if meets the criteria.
  Interventions: Drug: 131 I-Metaiodobenzylguanidine (131I-MIBG); Drug: Potassium iodide solution; Drug: G-CSF; Procedure: hematopoietic stem cell infusion

INTERVENTIONS:
Drug: 131 I-Metaiodobenzylguanidine (131I-MIBG) — Minimum dose of 10 mCi/kg and up to 18 mCi/kg maximum will be diluted in 25 ml of normal saline, and will be infused intravenously over 90-120 minutes.
  Other Names: 131I-MIBG
Drug: Potassium iodide solution — For the therapeutic MIBG administration, potassium iodide solution will be administered in a loading dose of 6mg/kg orally at least 8 hours prior to the MIBG injection, and then will be given at 1mg/kg/dose every 4 hours on days 0-6, then 1 mg/kg/day through day 45 post injection. The minimum dose of potassium iodide to be given is one drop, which equals 50 mg.
  Other Names: KI solution
Drug: G-CSF — It is recommended that patients with ANC less than 750 after MIBG infusion begin G-CSF 5 mcg/kg/day subcutaneously (or receive equivalent single dose of Neulasta every 14 days while neutropenic) until neutrophil recovery (generally >5000).
  Other Names: Neulasta
Procedure: hematopoietic stem cell infusion — The majority of patients on this protocol will have autologous PBSCs available. Allogeneic stem cells may be utilized in patients who has received a prior allogeneic transplant. The minimum quantity for peripheral blood stem cells is 1.5 x 106 CD34+ cells/kg (optimum > 2 x 106 CD34+ cells/kg). The minimum dose for bone marrow is 1.0 x 108 mononuclear cells/kg (optimum >2.0 x 108 mononuclear cells/kg). Infusion will be performed according to institutional guidelines.
  Other Names: HSCT

SUMMARY:
This is a best available therapy/compassionate use single institution study designed to determine the palliative benefit and toxicity of 131I-MIBG in patients with progressive neuroblastoma and metastatic pheochromocytoma who are not eligible for therapies of higher priority. Patients may receive a range of doses depending on stem cell availability and tumor involvement of bone marrow. Response rate, toxicity, and time to progression and death will be evaluated.

DETAILED DESCRIPTION:
Primary Objective is to provide access to therapy with 131I-MIBG for patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma.

Secondary Objective is to assess disease response to 131I-MIBG therapy for patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma.

Tertiary Objectives are to 1) gain more information about the toxicities of 131I-MIBG therapy; 2) assess improvement of symptoms, including pain and fatigue, for patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma who are receiving 131I-MIBG therapy.

* The therapeutic dose of 131I-MIBG will be based on the following:

  1. Minimum dose of 10 mCi/kg for patients without a stem cell source whose renal function is above the upper limit of normal but still meets eligibility criteria.
  2. Dose of 12 mCi/kg for patients without a stem cell source with normal renal function and meets other eligibility criteria.
  3. Dose of > 12 mCi/kg to 18 mCi/kg maximum at investigator's discretion for patients meeting eligibility criteria with stem cells available.
* A urinary catheter and intravenous fluids will be used for bladder protection, and potassium iodide solution for thyroid Protection.
* G-CSF is recommended for patients with ANC less than 750 after MIBG infusion.
* hematopoietic stem cell infusion is recommended for patients with grade 4 hematologic toxicity following 131I-MIBG therapy that continues to have an ANC <200 on G-CSF without signs of recovery for >2 weeks and any patient requiring platelet transfusion more than two times weekly for 4 consecutive weeks.
* Follow-up will be done until disease progression, death or other therapies are initiated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Relapsed/refractory neuroblastoma with original diagnosis based on tumor histopathology or elevated urine catecholamines with typical neuroblastoma cells in the bone marrow
  * Metastatic pheochromocytoma
* Age >1 year and able to cooperate with radiation safety restrictions during therapy period
* Karnofsky or Lansky performance status of ≥ 50%
* Life expectancy: ≥ at least 8 weeks
* Disease status: Failure to respond to standard therapy or development of progressive disease at any time.
* Disease must be evaluable by MIBG scan. A positive MIBG scan must be present within 8 weeks prior to study entry and subsequent to any intervening therapy. If the patient has only one MIBG positive lesion and that lesion was radiated, a biopsy must be done at least 4 weeks after radiation was completed and must show viable neuroblastoma.
* Stem Cells: Patients must have a hematopoietic stem cell product available for reinfusion after MIBG treatment at doses of > 12 mCi/kg.
* Have acceptable organ function as defined below within 7 days of enrollment:

  * Bone Marrow: ANC ≥750 X 109 /L and platelets ≥50,000 X 109 /L without transfusion if stem cells are not available (any ANC or platelet allowed if stem cells available)
  * Renal: Creatinine ≤3x upper limit of normal
  * Hepatic: Bilirubin ≤2x upper limit of normal; AST/ALT ≤10x upper limit of normal
  * Cardiac: Ejection fraction ≥45% on echocardiogram
  * Pulmonary: normal lung function as manifested by no dyspnea and/or oxygen saturation ≥ 88% on room air.
* Prior Therapy: Patients must have recovered from all acute toxicities (defined as CTCAE 4.0 ≤ grade 1) associated with any prior therapy, and:

  * Myelosuppressive chemotherapy: At least 2 weeks should have elapsed since any chemotherapy causing myelosuppression
  * Biologic (anti-neoplastic agent): At least 7 days should have elapsed since the completion of therapy with a biologic agent.
  * Monoclonal antibodies: At least 3 half-lives should have elapsed since therapy with a monoclonal antibody
  * Radiation therapy: Three-months should have elapsed in the case of completing radiation to any of the following fields: craniospinal, total abdominal, whole lung, total body irradiation). For all other sites of radiation, at least 2 weeks should have relapsed.
  * Cytokine therapy (e.g. G-CSF, GM-CSF, IL-6, IL-2): must be discontinued a minimum of 24 hours prior to MIBG therapy.
* Voluntary written informed consent

Exclusion Criteria:

* Patients with disease of any major organ system that would compromise their ability to withstand therapy.
* Because of the teratogenic potential of the study medication, no patients who are pregnant or lactating will be allowed. Patients of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus.
* Known allergy to any of the agents or their ingredients used in this study.
* Patients who are on hemodialysis
* Patients with untreated positive blood cultures or progressive infections as assessed by radiographic studies

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Number of patients who receive 131 I-MIBG. | 2 hours
  The number of patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma who receive access to 131 I-MIBG.

SECONDARY OUTCOMES:
Disease response | 1 year
  Disease response to 131 I-MIBG therapy in patients with relapsed/refractory neuroblastoma or metastatic pheochromocytoma. Disease response will be measured by Curie Score for patients with MIBG avid disease only or by both Currie Score and RECIST criteria for patients who have measureable disease in addition to MIBG avid disease. Disease response will be assessed at day 56 (+/- 14 days) and then every 3 months until 1-year post treatment, then every 6 months until progression, death or other therapy.
Incidence of hematologic toxicities | 1 year
  Evaluation of hematologic toxicities of 131I MIBG therapy. CBC with differential and platelet count will be obtained prior to study enrollment, on day 0 and then twice weekly until ANC>500/mm3 and platelet count >20,000 x 3 days without transfusion. Once that is achieved CBC will be then obtained on day 56 and then every 3 months until 1 year post treatment, then every 6 months until progression, death or other therapy. In addition, we will be looking at the percent of patient that require infusion of stem cell product for cytopenias.
Incidence of hepatic toxicities | 1 year
  ALT, AST, bilirubin will be obtained prior to study enrollment and then weekly until day 42, again on day 56 and then every 3 months until 1 year post treatment, then every 6 months until progression, death or other therapy
Incidence of Thyroid Toxicity | 1 year
  T4 and TSH will be obtained prior to study enrollment and again on day 56 and then every 3 months until 1 year post treatment, then every 6 months until progression, death or other therapy.
Improvement of pain symptoms | 56 days
  Assessment of pain will occur on day 0 of therapy, on the day of discharge and then weekly until day 42 and then again on day 56. The PedsQL Pediatric Pain Questionnaire will be used for assessment of pain in all patients. These questionnaires include both patient report and parent report, when appropriate.
Improvement of fatigue | 56 days
  Assessment of fatigue will occur on day 0 of therapy, on the day of discharge and then weekly until day 42 and then again on day 56. The PedsQL Multidimensional Fatigue Scale will be used for assessment of fatigue in all patients. These scales include both patient report and parent report, when appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Greengard, MD, Principal Investigator — University of Minnesota Department of Pediatrics
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT01850888/ICF_000.pdf